CLINICAL TRIAL: NCT03051477
Title: A Phase I Dose Escalating Trial of Mistletoe Extract in Patients With Advanced Solid Tumors
Brief Title: Trial of Mistletoe Extract in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Believe Big (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1681; IRB00090991 (Other: JHMIRB); Helixor (Other: Helixor Heilmittel GmbH & Co. KG.)
Record Dates: First submitted 2017-02-02; First posted 2017-02-13 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Helixor® M (Experimental): Advanced solid tumors
  Interventions: Drug: Helixor® M

INTERVENTIONS:
Drug: Helixor® M — 3-hour IV infusion on Monday, Wednesday, and Friday of each week.
  Other Names: Mistletoe extract

SUMMARY:
This study will seek to determine the safety and toxicity profile as well as the maximum tolerated dose of Helixor® M in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a Phase I study that consists of two phases: a dose escalation phase and an expansion phase. The dose escalation phase will be used to evaluate the safety and toxicity of Helixor® M (mistletoe extract). An accelerated titration design (ATD) will be utilized to determine the MTD. The expansion phase will be used to obtain preliminary efficacy data about Helixor® M.

ELIGIBILITY:
Any patients who have had any prior treatment with Mistletoe (injection or infusion) will not be eligible for this study.

Inclusion Criteria

* Patients with advanced solid tumors and have received first line standard systemic therapy with chemotherapy, immunotherapy, hormonal therapy or other standard treatments for metastatic disease. Patients must either have progressed, are refractory, have stable disease and/or removed from therapy due to toxicities. Patients beyond first line therapy that do not meet criteria may be considered on a case by case basis and allowed at discretion of PI.
* Patients with the presence of at least one measurable lesion as defined by RECIST 1.1 criteria for response assessment. Prostate cancer patients with bone disease only are eligible.
* Age >18 years.
* ECOG performance status 0-2
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below (without growth factor or transfusion support within 14 days prior to first dose of investigational product):

  * WBC ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 90,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 X ULN (patients with diagnosed Gilbert's Syndrome will not be excluded if their direct bilirubin is within normal institutional limits)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X ULN
  * Creatinine ≤1.5 x ULN OR creatinine clearance ≥ 50 mL/min/1.73 m2
* Female patient of childbearing potential has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible.
* Female patients enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from heterosexual activity throughout the study, starting with Visit 1 through 28 days after the last dose of study therapy. Approved contraceptive methods include for example; intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, female condoms with spermicide, or oral contraceptives. Spermicides alone are not an acceptable method of contraception.

  -- Male patients must agree to use an adequate method of contraception starting with the first dose of study drug through 28 days after the last dose of study therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patient with a known history or evidence of brain metastases.
* Patients who have had chemotherapy, radiation, hormonal, or biological cancer therapy within 28 days prior to the first dose of study drug excluding patients on long term hormonal therapies who have been on a stable dose for at least 3 months.
* Patient is currently participating or has participated in a study of an investigational agent or using an investigational device within 28 days of the first dose of study drug.
* Patients who have had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc), celiac plexus block, and biliary stent placement.
* Patient is expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Patient who has had prior treatment with Mistletoe.
* Patients who have received systemic corticosteroids within 28 days prior to the first dose of study drug. Note: Systemic steroid therapy is allowed for subjects on replacement therapy as long as prednisone ≤ 10 mg or its steroid equivalent.
* Patients who have received systemic NSAID therapy within 14 days prior to the first dose of study drug.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Mistletoe.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Presence of ≥ CTCAE grade 2 toxicity (except peripheral neuropathy and ototoxicity, which are excluded if ≥ CTCAE grade 3) due to prior cancer therapy.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis, multiple sclerosis). History of Grave's disease on stable thyroid hormone replacement for at least 1 year is allowed.
* Patients with a known history of HIV, hepatitis B, hepatitis C, or tuberculosis infection. Patients with a history of cleared hepatitis C (undetectable viral loads) are allowed.
* Women with a positive pregnancy test on enrollment or prior to investigational product administration
* Women who are pregnant or breastfeeding.
* Sexually active fertile men not using effective birth control if their partners are of child bearing potential.
* Patient is unwilling or unable to comply with study procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing toxicities | 3 years
  Number of participants who experience side effects
Maximum tolerated dose (MTD) | 2 years
  The highest dose that does not cause unacceptable side effects

SECONDARY OUTCOMES:
Tumor marker kinetics | 3 years
  Changes in disease specific bio markers: analyzed as percent change and presented in a waterfall plot of response.

CONTACTS AND LOCATIONS:
Overall Officials: Channing Paller, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No